CLINICAL TRIAL: NCT00409968
Title: A Biomarker-Integrated Study in Chemorefractory Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: BATTLE Program: Umbrella Protocol for Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2005-0823; W81XWH-06-1-0303 (Other: U.S. Department of Defense); NCI-2018-01767 (Registry Identifier: CTRP ID)
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non Small Cell Lung Cancer; BATTLE Program; Umbrella Trial; Tumor Biopsy; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A sample of your tumor tissue will be collected for biomarker analysis, and based on the results, you will be assigned to one of four phase II studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening Study: Screening study to find out if Patients with non-small cell lung cancer (NSCLC) that has spread to other parts of the body are eligible to take part in 1 of 4 different research studies.
  Interventions: Procedure: Tumor Biopsy

INTERVENTIONS:
Procedure: Tumor Biopsy — A sample of tumor tissue will be collected by either a CT-guided core biopsy, bronchoscopy, or other type of biopsy (such as subcutaneous, cutaneous, or lymph node).

SUMMARY:
This trial is referred to as the "umbrella trial". The BATTLE program consists of this umbrella trial plus four phase II protocols into which the umbrella patients are enrolled. Patients will first enroll in the BATTLE umbrella trial and undergo a tumor biomarker analysis that will be used to assign them to one of the four phase II studies. All patients enrolled in one of the phase II BATTLE protocols must be enrolled in this protocol.

DETAILED DESCRIPTION:
This study is the "umbrella" or screening study in a group of 5 studies known as the BATTLE (Biomarker-integrated Approaches of Targeted Therapy of Lung Cancer Elimination) program. In order to participate in one of the research studies, you must first agree to take part in this screening study, which will be used to determine if you are eligible. After participating in this study, you may be assigned to a study that is using an investigational drug. The investigational drug(s) to be used in each of the 4 studies are not approved by the Food and Drug Administration (FDA) for commercial use in this setting; however, the FDA has permitted its use in these research studies.

If you agree to participate in this screening study, your complete medical history (including smoking history) will be recorded and you will have a physical exam, including measurement of vital signs (blood pressure, pulse, temperature, and breathing rate), height, and weight. You will have blood (about 2 teaspoons) drawn for routine tests. You will also have blood (about 1-2 tablespoons) drawn to check your blood clotting function, thyroid function, and lipid (fat) levels. You will have a urine test, a performance status evaluation (questions about your ability to perform everyday activities), and an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).

Your tumor will be evaluated by chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans to evaluate the status of the disease. You will have a brain MRI. Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test before receiving the study drug.

A sample of your tumor tissue will be collected for biomarker analysis. If your tumor tissue cannot be reached, you will not be able to participate in this research study. To collect a tumor biopsy, you will have either a CT-guided core biopsy, bronchoscopy, or other type of biopsy (such as subcutaneous, cutaneous, or lymph node). You will be asked to stop taking any medication that affects blood-clotting (such as aspirin or coumadin) before the biopsy procedure.

For the cutaneous (skin) biopsy, you will be given a local anesthetic by either a spray or shot to numb your skin. A small cut will be made to remove all or a piece of the affected skin.

For the CT-guided core biopsy of the lung, subcutaneous, and/or lymph node biopsy, a tissue sample is withdrawn from an organ or suspected tumor mass using a very thin needle and a syringe. The needle is guided while being viewed by the physician on a CT scan. Any site that can be safely biopsied will be considered for the collection of tissue. Sites not commonly biopsied include kidneys, adrenal glands, and brain.

For the bronchoscopy, you will be given drugs to relax, and then a local anesthetic will be sprayed into your nose and throat to numb those areas. A slim, flexible tube with a light will be placed through your nose or mouth and into your lungs. A small brush will be fed through the tube and into your lungs. The brush will gently scrape off a sample of lung tissue. Tweezers will then be fed through the tube to collect the tissue samples (biopsy). A small amount of water will be sprayed into your lungs and then suctioned out through the tube to collect tissue samples and mucous samples.

For the CT-guided core biopsy or bronchoscopy, you should not take any medications by mouth or have any solid food for at least 6 hours before the procedure. You also should not have any liquids 2 hours before the procedure.

If you are eligible to take part in this study, you will be assigned to 1 of the 4 research studies based on the results of your tumor analysis. You will be asked to read and sign a separate informed consent to take part in one of the research studies.

You have the right to leave the study at any time. If you choose to stop participating in this study, you should contact the study chair and/or research nurse. Your doctor may decide to take you off this study if your medical condition gets worse and/or you are unable to comply with study requirements.

This is an investigational study. Up to 250 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration
2. The patient has a diagnosis of either stage IIIB, stage IV, or advanced, incurable NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen. (Patients who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in study).
3. The patient has uni-dimensionally measurable NSCLC.
4. Karnofsky performance status >/= 60 or ECOG performance status 0-2
5. The patient has biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, WBC >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 X the upper limit of normal, and alkaline phosphatase, AST or ALT </= 2.5 X the upper limit of normal.
8. The patient has adequate renal function as defined by a serum creatinine level </= 1.5 mg/dL or a calculated creatinine clearance of >/= 60cc/minute.
9. The patient has PT < 1.5 x upper limit of normal
10. If patient has brain metastasis, they must have been stable (treated or asymptomatic) for at least 4 weeks after radiation if treated with radiation and not have used steroids for at least 1 week. Re-imaging performed after 2 weeks, upon completion of radiation therapy.
11. The patient is >/= 18 years of age.
12. The patient has signed informed consent.
13. The patient is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are exempt from exclusion.
14. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months,who have not had tubal ligation or bilateral oophorectomy.Should a woman become pregnant or suspect that she is pregnant while participating in this study,she should inform her treating physician immediately.The patient,if a man,agrees to use effective contraception or abstinence.
15. Subject must be considered legally capable of providing his or her own consent for participation in this study.

Exclusion Criteria:

1. The patient has received prior investigational therapy, chemotherapy, surgery, or radiotherapy within 4 weeks of initiating study drug
2. The patient has undergone prior thoracic or abdominal surgery within 28 days of study entry, excluding prior diagnostic biopsy.
3. The patient has received radiation therapy to the measurable tumor within 6 months. Patients are allowed to have local irradiation for the management of tumor-related symptoms (bones, brain). However, if a patient has active new disease growing in the previously irradiated site, the patient will be eligible to participate in the study.
4. The patient has a significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure (New York Heart Association Functional Classification class II or worse), recent myocardial infarction within 3 months, unstable angina, active infection (i.e. currently treated with antibiotics), uncontrolled hypertension). Patients with controlled diabetes will be allowed. Patient must be able to undergo procedure for tissue acquisition.
5. The patient has uncontrolled seizure disorder, active neurologic disease, or neuropathy >/= grade 2. Patients with meningeal or CNS involvement by tumor are eligible for the study if the above exclusion criteria are not met.
6. The patient is pregnant (confirmed by serum Beta-HCG if applicable) or is breastfeeding.
7. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.
8. The patient is actively taking herbal remedies or over-the-counter biologics (e.g., shark cartilage, high dose antioxidants).
9. Patients will be allowed to have prior biologic (i.e. VEGF, EGFR, etc.) therapy. However, the patient will be excluded from a given study if he/she has received the same therapy as the clinical trial (i.e. If a patient has been previously treated with bevacizumab, they are allowed to enroll in any of the 4 studies. If a patient has been previously treated with erlotinib, they are excluded from the clinical trials with erlotinib). In addition, if a patient has been previously treated with gefitinib (Iressa), they are excluded from the clinical trials with erlotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer (NSCLC) that has spread to other parts of the body.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2006-11-27 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Biomarker Profile Assessment (before randomized allocation to research study) | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Vali Papadimitrakopoulou, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Seguin L, Kato S, Franovic A, Camargo MF, Lesperance J, Elliott KC, Yebra M, Mielgo A, Lowy AM, Husain H, Cascone T, Diao L, Wang J, Wistuba II, Heymach JV, Lippman SM, Desgrosellier JS, Anand S, Weis SM, Cheresh DA. An integrin beta(3)-KRAS-RalB complex drives tumour stemness and resistance to EGFR inhibition. Nat Cell Biol. 2014 May;16(5):457-68. doi: 10.1038/ncb2953. Epub 2014 Apr 20. PMID 24747441
- [Derived] Tam AL, Kim ES, Lee JJ, Ensor JE, Hicks ME, Tang X, Blumenschein GR, Alden CM, Erasmus JJ, Tsao A, Lippman SM, Hong WK, Wistuba II, Gupta S. Feasibility of image-guided transthoracic core-needle biopsy in the BATTLE lung trial. J Thorac Oncol. 2013 Apr;8(4):436-42. doi: 10.1097/JTO.0b013e318287c91e. PMID 23442309
- [Derived] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org